CLINICAL TRIAL: NCT04776161
Title: Using Cues and Rewards in Patients With Arthritis and Rheumatic Disease
Brief Title: Medication Adherence Patterns in Rheumatic Diseases: A Behavioral Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Candace Hillary Feldman, MD, Assistant Professor, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 2020P003826; P30AG064199-01 (NIH)
Record Dates: First submitted 2021-02-23; First posted 2021-03-01 (Actual); Results first posted 2023-10-04 (Actual); Last update posted 2023-10-04 (Actual); Status verified 2023-09

CONDITIONS: Rheumatic Diseases; Gout; Adherence, Medication; Lupus Erythematosus, Systemic
MeSH Terms: conditions — Rheumatic Diseases; Gout; Medication Adherence; Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): Patients in the control arm will not receive any intervention (but will receive electronic pill bottles to monitor their adherence).
- Cue-Reward Intervention (Experimental): Patients in this intervention arm will choose an event-based cue and receive reminder text messages reminding them of their cue. Additionally, a donation will be made to a local charity every time they take their medication.
  Interventions: Behavioral: Cue-Reward Intervention
- Cue-Reward Intervention with possible intensification. (Experimental): Patients in this intervention arm will choose an event-based cue. Additionally, a donation will be made to a local charity every time they take their medication. Those who show no improvement in adherence after 6 weeks will start receiving reminder text messages reminding them of their cue.
  Interventions: Behavioral: Cue-Reward Intervention with possible intensification

INTERVENTIONS:
Behavioral: Cue-Reward Intervention — Patients in the first intervention arm will participate in a goal-setting exercise during which they will identify which habit they want to link their medication-taking to. Patients will also receive text messages reminding them of the habit they decided to link to their medication-taking.
  Finally, patients will also select a charity to which a donation will be made every time the bottle is opened. The research team will donate $0.50 every day that the patient takes their medication as prescribed. A research assistant will place a sticker with the charity logo under the pill bottle cap so that the patient is reminded of the donation every time they take the medication. Additionally, the patient will receive texts every 4 days summarizing how much money was donated on their behalf.
  Arms: Cue-Reward Intervention
Behavioral: Cue-Reward Intervention with possible intensification — Patients in the second intervention arm will participate in a goal-setting exercise during which they will identify which habit they want to link their medication-taking to. Finally, patients will also select a charity to which a donation will be made every time the bottle is opened. The research team will donate $0.50 every day that the patient takes their medication as prescribed. A research assistant will place a sticker with the charity logo under the pill bottle cap so that the patient is reminded of the donation every time they take the medication. Additionally, the patient will receive texts every 4 days summarizing how much money was donated on their behalf.
  After 6 weeks, patients who demonstrate an adherence under 80% to study medications (as measured by the electronic pill bottle) will begin receiving text messages reminding them of their selected cue.
  Arms: Cue-Reward Intervention with possible intensification.

SUMMARY:
Non-adherence to evidence-based prescription medications results in preventable morbidity and mortality for middle-aged and older adults. Taking medications intended for daily use, like those to prevent or treat chronic conditions, is a repetitive action that has great similarity with other behaviors that must be performed consistently, such as regular exercise, healthy eating, and hand washing. In these cases, people who act consistently do so out of habit. The "repetition-cue-reward" model proposes that habit formation has three central components: behavioral repetition, associated context cues, and rewards. This model has obvious applicability to the daily repetitive activity of medication-taking but has not been tested for this behavior nor adapted as an intervention for patients in real-world care settings.

The goal of this pilot study is to evaluate the feasibility and effectiveness of using the repetition-cue-reward model of healthy habit formation to improve medication adherence in patients with arthritis and other rheumatic diseases.

DETAILED DESCRIPTION:
Non-adherence to evidence-based prescription medications results in preventable morbidity and mortality for middle-aged and older adults. Taking medications intended for daily use, like those to prevent or treat chronic conditions, is a repetitive action that has great similarity with other behaviors that must be performed consistently, such as regular exercise, healthy eating, and hand washing. In these cases, people who act consistently do so out of habit. The "repetition-cue-reward" model proposes that habit formation has three central components: behavioral repetition, associated context cues, and rewards. This model has obvious applicability to the daily repetitive activity of medication-taking but has not been tested for this behavior nor adapted as an intervention for patients in real-world care settings.

The goal of this pilot study is to evaluate the feasibility and effectiveness of using the repetition-cue-reward model of healthy habit formation to improve medication adherence in patients with arthritis and other rheumatic diseases.

This pilot study will be a 3-arm parallel randomized pragmatic trial comparing medication adherence for adults over 18 years old with arthritis, lupus, or gout who are prescribed 1-3 daily oral medications for this disease. Participants will be randomized to one of three arms for the duration of the study period. Patients in the first intervention arm will choose an event-based cue and receive daily reminder text messages reminding them of their cue. Patients in the second intervention arm will start by establishing their cue and having the donation made, but only those who show no improvement in adherence after 6 weeks will start receiving the text messages. In both interventions arms, a donation will be made to a local charity every time they take their medication. Patients in the control arm will not receive any intervention (but will receive pill bottles to monitor their adherence). Our outcomes of interest will be medication adherence, as measured by electronic pill bottles.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking patients
* receiving their care at a Brigham and Women's Hospital-affiliated rheumatology practice
* >=18 years of age
* with rheumatoid arthritis (RA), systemic lupus erythematosus (SLE), or gout
* prescribed >=1 oral medication for this disease for >=4 months.
* for patients with gout, had a uric acid level checked in the prior 18 months and the most recent level is >6.
* for patients with SLE, their most recent c-reactive protein level collected in the past 18 months must be >10.
* currently have a smartphone with a data plan or WiFi at home
* willing and able to set up the platform and adhere to study procedures
* either not currently using a pillbox or willing to use electronic pill bottles (EDMs) for diabetes medications for the duration of the study

Exclusion Criteria:

* Pregnant women
* Incarcerated individuals

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2021-08-02 (Actual); Primary Completion 2022-09-27 (Actual); Study Completion 2022-11-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Candace H Feldman, MD, ScD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Fontanet CP, Choudhry NK, Wood W, Robertson T, Haff N, Oran R, Sears ES, Kim E, Hanken K, Barlev RA, Lauffenburger JC, Feldman CH. Randomised controlled trial targeting habit formation to improve medication adherence to daily oral medications in patients with gout. BMJ Open. 2021 Nov 24;11(11):e055930. doi: 10.1136/bmjopen-2021-055930. PMID 34819291

RESULTS

PARTICIPANT FLOW:
Groups:
- Non-adaptive Intervention: Patients in this intervention arm will choose an event-based cue and receive reminder text messages reminding them of their cue. Additionally, a donation will be made to a local charity every time they take their medication.
  Cue-Reward Intervention: Patients in the first intervention arm will participate in a goal-setting exercise during which they will identify which habit they want to link their medication-taking to. Patients will also receive text messages reminding them of the habit they decided to link to their medication-taking.
  Finally, patients will also select a charity to which a donation will be made every time the bottle is opened. The research team will donate $0.50 every day that the patient takes their medication as prescribed. A research assistant will place a sticker with the charity logo under the pill bottle cap so that the patient is reminded of the donation every time they take the medication. Additionally, the patient will receive texts every 4 days summarizing how much money was donated on their behalf.
- Adaptive Intervention: Patients in this intervention arm will choose an event-based cue. Additionally, a donation will be made to a local charity every time they take their medication. Those who show no improvement in adherence after 6 weeks will start receiving reminder text messages reminding them of their cue.
  Cue-Reward Intervention with possible intensification: Patients in the second intervention arm will participate in a goal-setting exercise during which they will identify which habit they want to link their medication-taking to. Finally, patients will also select a charity to which a donation will be made every time the bottle is opened. The research team will donate $0.50 every day that the patient takes their medication as prescribed. A research assistant will place a sticker with the charity logo under the pill bottle cap so that the patient is reminded of the donation every time they take the medication. Additionally, the patient will receive texts every 4 days summarizing how much money was donated on their behalf.
  After 6 weeks, patients who demonstrate an adherence under 80% to study medications (as measured by the electronic pill bottle) will begin receiving text messages reminding them of their selected cue.
Period: Overall Study
Arm/Group | Control | Non-adaptive Intervention | Adaptive Intervention
Started | 19 | 21 | 22
Completed | 17 | 17 | 18
Not Completed | 2 | 4 | 4
Not completed — Withdrew after randomization but prior to intervention | 1 | 3 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 1
Not completed — Adverse Event | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: We consented and randomized 62 participants in total (see Results Participant Flow).
  However, 6 participants never started the trial, so they are not included in the Baseline Analysis Population. Thus, the baseline population represented here are the 56 participants who consented and initiated the trial. Those 6 participants are reflected in the Results Participant Flow under withdrawal reason "withdrew after randomization but prior to intervention."
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Non-adaptive Intervention | Adaptive Intervention | Total
Number analyzed (Participants) | 18 | 18 | 20 | 56
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.8 (12.5) | 50.7 (12.4) | 60.2 (11.8) | 55.6 (12.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 5 | 11
  Male | 16 | 14 | 15 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 1 | 4
  Not Hispanic or Latino | 17 | 16 | 19 | 52
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 3 | 4 | 2 | 9
  White | 14 | 13 | 17 | 44
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1 | 2
Uric Acid Level [Mean (Standard Deviation); unit: mg/dL] — Mean (SD) baseline uric acid level
  mg/dL | 7.07 (0.90) | 7.92 (2.31) | 7.43 (1.06) | 7.47 (1.55)

OUTCOME MEASURES:

1. Primary Outcome: Rate of Medication Adherence
Description: Medication adherence will be measured as the percentage of times a patient opened the electronic pill bottle out of the number of doses prescribed for each bottle in each day, averaged across the study medications and over follow-up.
Time Frame: 18 weeks
Measure: Mean (Standard Deviation); unit: percentage of doses taken
Arm/Group | Control | Non-adaptive Intervention | Adaptive Intervention
Number analyzed (Participants) | 18 | 18 | 20
percentage of doses taken | 0.76 (0.26) | 0.79 (0.23) | 0.83 (0.18)
Statistical Analysis 1: Comparison: Control vs Non-adaptive Intervention; Test type: Superiority; p = 0.78, Generalized linear models; Adjusted for age, sex, race; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.16 to 0.12]
Statistical Analysis 2: Comparison: Control vs Adaptive Intervention; Test type: Superiority; p = 0.79, Generalized linear models; Adjusted for age, sex, race; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.10 to 0.13]

2. Secondary Outcome: Change in Uric Acid Level From Baseline
Description: Change in uric acid level from baseline
Time Frame: 18 weeks
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)
Arm/Group | Control | Non-adaptive Intervention | Adaptive Intervention
Number analyzed (Participants) | 18 | 18 | 20
milligrams per deciliter (mg/dL) | -1.21 (1.31) | -1.13 (1.66) | -0.55 (1.88)
Statistical Analysis 1: Comparison: Control vs Non-adaptive Intervention; Test type: Superiority; p = 0.22, Generalized linear models; Adjusted for age, sex, race and baseline uric acid level; Mean Difference (Final Values) = 0.47, 95% CI 2-sided [-0.28 to 1.22]
Statistical Analysis 2: Comparison: Control vs Adaptive Intervention; Test type: Superiority; p = 0.24, Generalized linear models; Adjusted for age, sex, race and baseline uric acid level; Mean Difference (Final Values) = 0.47, 95% CI 2-sided [-0.33 to 1.26]

ADVERSE EVENTS:
Time Frame: Adverse events were collected through the entire trial period of 18 weeks.
Arm/Group | Control | Non-adaptive Intervention | Adaptive Intervention
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/18 | 0/20
Serious Adverse Events (participants affected / at risk) | 1/18 | 2/18 | 3/20
Other Adverse Events (participants affected / at risk) | 0/18 | 0/18 | 0/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=18) | Non-adaptive Intervention (N=18) | Adaptive Intervention (N=20)
Hospitalization for congestive heart failure (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Hospitalization for fall-related complications (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Kidney transplant (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Appendectomy (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Hospitalization for secondary hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1)
Hospitalization for colostomy leak (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Ileostomy reversal (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2022-10-10): https://cdn.clinicaltrials.gov/large-docs/61/NCT04776161/Prot_000.pdf
  • Statistical Analysis Plan (2022-12-16): https://cdn.clinicaltrials.gov/large-docs/61/NCT04776161/SAP_002.pdf
  • Informed Consent Form (2021-07-12): https://cdn.clinicaltrials.gov/large-docs/61/NCT04776161/ICF_001.pdf